CLINICAL TRIAL: NCT02391415
Title: Phase II Double-blind, Randomized, Controlled Study to Evaluate Safety and Immunogenicity of VPM1002 Compared With BCG in HIV-exposed and HIV-unexposed, BCG-naive Newborn Infants
Brief Title: Study to Evaluate the Safety and Immunogenicity of VPM1002 in Comparison With BCG in HIV-exposed/-Unexposed Newborn Infants in South Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: Serum Life Science Europe GmbH (Industry); Triclinium Clinical Trial Project Management (Unknown); Children's Infectious Diseases Clinical Research Unit (KID-CRU) (Unknown); Desmond Tutu TB Centre (Other); The Respiratory and Meningeal Pathogens Research Unit (RMPRU) (Unknown); South African Tuberculosis Vaccine Initiative (Other); University of Stellenbosch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VPM1002-ZA-2.13TB; DOH-27-1114-4798 (Other: NHREC)
Record Dates: First submitted 2015-03-05; First posted 2015-03-18 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- HIV-unexposed infants VPM1002 (Experimental): HIV-unexposed infants vaccinated with VPM1002
  Interventions: Biological: VPM1002
- HIV-unexposed infants BCG (Active Comparator): HIV-unexposed infants vaccinated with BCG
  Interventions: Biological: BCG
- HIV-unexposed infants VPM1002(Hyg+) (Experimental): HIV-unexposed infants vaccinated with VPM1002(Hyg+)
  Interventions: Biological: VPM1002(Hyg+)
- HIV-exposed infants BCG (Active Comparator): HIV-exposed infants vaccinated with BCG
  Interventions: Biological: BCG
- HIV-exposed infants VPM1002 (Experimental): HIV-exposed infants vaccinated with VPM1002
  Interventions: Biological: VPM1002

INTERVENTIONS:
Biological: VPM1002 — Tuberculosis vaccine
  Other Names: recombinant BCG for TB
  Arms: HIV-exposed infants VPM1002; HIV-unexposed infants VPM1002
Biological: BCG — commercially available live vaccine BCG
  Arms: HIV-exposed infants BCG; HIV-unexposed infants BCG
Biological: VPM1002(Hyg+) — Tuberculosis vaccine
  Other Names: recombinant BCG for TB
  Arms: HIV-unexposed infants VPM1002(Hyg+)

SUMMARY:
Goal of Serum Institute of India Limited (SIIL) is the development of a recombinant urease C-deficient listeriolysin expressing BCG vaccine strain (VPM1002) as a safe, well tolerated and efficacious vaccine against tuberculosis (TB) for residents in endemic areas and persons at risk in non-endemic areas. The new vaccine should be at least as potent as the current strain and should be safer than BCG.

The preceding phase-IIa trial was the first investigation of VPM1002 in newborn infants in a high burden setting in South Africa. The vaccination of HIV-unexposed infants with VPM1002 indicated again safety, tolerability and immunogenicity sufficient to proceed in HIV-exposed infants.

The current study is a multiple site trial in South Africa to evaluate safety and immunogenicity in HIV-unexposed and -exposed newborn infants.

ELIGIBILITY:
Inclusion Criteria:

Maternal:

1. The infant's mother must be aged 18 years or older at screening.
2. The infant's mother must be able and willing to comply with the study protocol, available and willing to allow her child to complete all the study assessments and must have signed an Informed Consent form that has been approved by all relevant Ethics Committee/s.
3. The infant's mother must not have any symptoms or signs of active TB as indicated by history of cough for more than two weeks, fever, weight loss, breathlessness, chest pain, blood in sputum, night sweats and loss of appetite
4. The infant's mother should not be planning to relocate from the research site area and should be reachable by phone during the whole study period i.e. for the 12 months on-study period as well as the 24 month structured medical surveillance period.
5. For HIV-unexposed group: The infant's mother must test negative for HIV-1 (ELISA 4th generation) within the period from 2 weeks prior to the infant's birth to vaccination of the infant with the investigational product.

   For the HIV-exposed group: The infant's mother must test positive for HIV-1 (ELISA 4th generation) within the period from 2 weeks prior to the infant's birth to vaccination of the infant with the investigational product. The infant's mother must have enrolled for standard antiretroviral therapy (ART) at least 3 months before the participating infant's birth and must have a viral load at screening below 1000 copies/ml. The use of ART, including combination antiretroviral therapy (cART) and preventive mother to child transmission (PMTCT) must be documented. CD4+ T cell count and HIV viral load must be documented.
6. The infant's mother must test negative for Hepatitis B and syphilis serology at screening.
7. The infant's mother should have no history or evidence of diabetes mellitus.
8. No participation of the infant's mother in a clinical trial within 3 months prior to the birth of the participating infant. In addition, if breast-feeding, no participation in another clinical trial during the 12 months of the current study.
9. The infant's mother must have no known history of immunodeficiency, except for HIV.

Infant:

1. Healthy male or female newborn infants aged 0 to 12 days.
2. Infants must have a birth weight of 2500 - 4200 g and an Apgar score of > 7 at 5 minutes or earlier.
3. No eczema or other significant skin lesion or infection at the intended injection site.
4. No routine BCG vaccination administered (as per vaccination record)
5. Infants must receive Oral Polio Vaccine as part of the routine South African Expanded Programme on Immunisation (EPI) Childhood Immunisation schedule, and must adhere to the subsequent EPI schedule for the entire study period, except for the BCG vaccination at birth.
6. No participation of the infant in another clinical trial before study vaccination and during the 12 months of the current study.

Exclusion Criteria:

Maternal:

1. Known presence of any person in the household of the mother and newborn infant, or any recent visitor to the household with recently diagnosed, active tuberculosis disease (within last 3 months).
2. Treatment of the mother with blood products in the 6 months prior to or during the birth of the participating infant.
3. For the HIV-unexposed group: Positive test for HIV-1 either during the current pregnancy or at screening.

   For the HIV-exposed group: Negative test for HIV-1 either during the current pregnancy or at screening.
4. Presence of signs or symptoms of any reported acute infectious disease at the time of screening.
5. Any reported or suspected substance abuse.

Infant:

1. History or evidence of any systemic disease on physical examination or any acute, chronic or intercurrent illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.

   Note: Neonatal jaundice not considered clinically significant by the investigator is not an exclusion.
2. Fever within the period post birth and prior to dosing. For the purposes of this protocol, fever in the infant will be defined as an axillary body temperature > 38.0°C measured by digital thermometer on at least 2 occasions not less than 6 hours apart.
3. Hypothermia within the period post birth and prior to dosing. For the purposes of this protocol, hypothermia in the infant will be defined as an axillary body temperature < 36.0°C measured by digital thermometer on at least 2 occasions not less than 6 hours apart.
4. Clinically suspected newborn sepsis.
5. Any malignant condition.
6. Any severe congenital malformation.
7. Concomitant treatment with medication that may significantly affect immune function (e.g. systemic corticoids, immunosuppressive drugs) before study vaccination. Antibiotics given before study vaccination would further constitute exclusion.
8. Treatment of the infant with blood products.

Max Age: 12 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 416 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The difference between the VPM1002 and BCG vaccination groups in the incidence of grade 3 and 4 adverse drug reactions and IMP-related ipsilateral or generalised lymphadenopathy of 10mm or greater (diameter). | up to 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- South Africa (4):
  - Children's Infectious Diseases Clinical Research Unit, Tygerberg Hospital, Cape Town
  - Desmond Tutu TB Centre, Cape Town
  - South African Tuberculosis Vaccine Initiative, Cape Town
  - The Respiratory and Meningeal Pathogens Reserach Unit, Johannesburg

REFERENCES:
- [Derived] Cotton MF, Madhi SA, Luabeya AK, Tameris M, Hesseling AC, Shenje J, Schoeman E, Hatherill M, Desai S, Kapse D, Bruckner S, Koen A, Jose L, Moultrie A, Bhikha S, Walzl G, Gutschmidt A, Kotze LA, Allies DL, Loxton AG, Shaligram U, Abraham M, Johnstone H, Grode L, Kaufmann SHE, Kulkarni PS. Safety and immunogenicity of VPM1002 versus BCG in South African newborn babies: a randomised, phase 2 non-inferiority double-blind controlled trial. Lancet Infect Dis. 2022 Oct;22(10):1472-1483. doi: 10.1016/S1473-3099(22)00222-5. Epub 2022 Jun 27. PMID 35772447